CLINICAL TRIAL: NCT02283957
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy and Safety of CNTX-4975 in Subjects With Painful Intermetatarsal Neuroma (Morton's Neuroma)
Brief Title: A Study to Evaluate the Efficacy and Safety of CNTX-4975 in Subjects With Painful Intermetatarsal Neuroma (Morton's Neuroma)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centrexion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4975-MN-202
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Painful Intermetatarsal Neuroma (Morton's Neuroma)
MeSH Terms: conditions — Morton Neuroma | interventions — CNTX-4975

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 2 mL injection of 200 µg of CNTX-4975 (Experimental): Single dose, 2 mL
  Interventions: Drug: CNTX-4975
- 2 mL injection of 600 µg of CNTX-4975 (Experimental): Single dose, 2 mL
  Interventions: Drug: CNTX-4975
- 2 mL injection of placebo (Placebo Comparator): Single dose, 2 mL
  Interventions: Other: Placebo
- 2 mL injection of 25 µg of CNTX-4975 (Experimental): Single dose, 2 mL
  Interventions: Drug: CNTX-4975

INTERVENTIONS:
Drug: CNTX-4975
  Arms: 2 mL injection of 200 µg of CNTX-4975; 2 mL injection of 25 µg of CNTX-4975; 2 mL injection of 600 µg of CNTX-4975
Other: Placebo
  Arms: 2 mL injection of placebo

SUMMARY:
Study 4975-MN-202 is a double-blind, placebo-controlled, parallel group, single-injection study in which subjects will be randomized to receive three doses of CNTX-4975 or placebo injected into the intermetatarsal space around a Morton's neuroma. The injection of study medication will be administered by ultrasound-guided needle placement following ankle block anesthesia. The study staff will telephone subjects at Week 1 postinjection and subjects will return to the clinic postinjection at Weeks 2, 4, 8, and 12 for study assessments.

ELIGIBILITY:
Inclusion criteria:

1. Male or female aged >18 years at the time of the Screening Visit.
2. Pain associated with intermetatarsal neuroma (Morton's neuroma) for a minimum of 3 months prior to Screening.
3. Diagnosis of Morton's neuroma, confirmed by evidence of focal tenderness and pain in the distal third intermetatarsal space, AND either

   * Presence of neuroma on ultrasound, or
   * Elicitation of Mulder's sign or a positive Gauthier's test.
4. A mean neuroma foot pain score of 4 or greater during the 7 days prior to dosing (NPRS, 0-10) as rated daily at bedtime (9:00 PM ± 3 hours) for average pain with walking in the last 24-hours. At least 5 of 7 scores during the week prior to dosing must be recorded.
5. Tried conservative treatment with analgesics (acetaminophen or nonsteroidal anti-inflammatory drugs) and non-pharmacologic therapy (such as wide shoes, orthotics, and/or arch supports) without complete success.
6. Female not of childbearing potential, defined as post-menopausal for at least 1 year, or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), or practicing one of the following medically acceptable methods of birth control throughout the study period:

   * Hormonal methods such as oral, implantable, injectable, or transdermal contraceptives for a minimum of 1 full cycle (based on the subject's usual menstrual cycle period) before investigational product (IP) administration.
   * Total abstinence from sexual intercourse since the last menses before IP administration.
   * Intrauterine device.
   * Double barrier method (condoms, sponge, diaphragm, with spermicidal jellies or cream).
7. Willing and able to understand the study requirements, abide by the study restrictions, complete the study procedures, pain scales, and daily IWRS/IVRS entries, and to communicate meaningfully with the study personnel.
8. Signed an Informed Consent Form approved by the Institutional Review Board.
9. Subject agrees to take only the rescue medications for neuroma foot pain from the time of screening through study completion, and agrees to discontinue all topical medications for neuroma pain after Screening.

Exclusion criteria:

1. Clinically significant bursitis in either foot.
2. The subject has more than one painful intermetatarsal neuroma in the affected foot which, in the opinion of the Investigator, would interfere with evaluation of the symptoms and functional limitations that arise from the intermetatarsal neuroma in the affected foot.
3. Radiography within 6 months of the Treatment Visit (Day 1) to exclude musculoskeletal pathology must be performed, to include any osseous abnormality such as stress fracture, osteophyte, tumor, or cyst in the bones or toes adjacent to the third inter-metatarsal space or any significant evidence of arthritis in the joints of the 3rd and 4th metatarsal-phalangeal joints or inter-phalangeal joints of the 3rd and 4th toes.
4. Previous neurectomy in the same nerve.
5. Any painful condition or prior surgery on the affected ankle or foot, which, in the judgment of the investigator, might adversely impact the interpretation of study data.
6. Other painful foot pathology (e.g., bunion, hammertoe, plantar fasciitis etc.) or evidence of clinically meaningful ischemia which, in the judgment of the investigator and the medical monitor, would interfere with evaluation of the symptoms and functional limitations that arise from the intermetatarsal neuroma.
7. Other chronic pain anywhere in the body that is greater than or equal to the intensity of foot pain from intermetatarsal neuroma.
8. Signs of arterial insufficiency in the feet, including clinically meaningful edema.
9. Current use of opioids for any condition.
10. Corticosteroid injection in the affected foot within 30 days of Screening.
11. History of clearly documented allergic reaction to local anesthetics or capsaicin.
12. Prior use of injection with a sclerosing agent, such as alcohol or phenol, in the affected foot for Morton's neuroma.
13. Presence of any medical condition or unstable health status that, in the judgment of the investigator, might adversely impact the conduct of the study or resulting data, including chronic conditions that are likely to alter the rate of healing or are likely to result in safety complications unrelated to the study medication, such as uncontrolled diabetes mellitus or vascular disease.
14. Regular use of anticoagulant blood thinners (except low-dose aspirin or Plavix which are allowed).
15. Active cutaneous disease at the anticipated site of study drug injection that would prevent the safe administration of study drug.
16. Ulcer or open wound anywhere on the affected foot.
17. Clinically significant abnormal laboratory result at the Screening Visit (in the opinion of the investigator).
18. Has diabetic neuropathy or other peripheral neuropathy in the affected foot.
19. Use of an investigational medication in the 30 days prior to the current study or scheduled to receive such an agent while participating in the current study.
20. Prior participation in an ALGRX-4975 or CNTX-4975 study.
21. Has a history of substance use disorder within the previous year as defined by the Diagnostic and Statistical Manual for Mental Health Disorders, fifth edition, has current evidence for a substance use disorder, is receiving medicinal treatment for drug abuse, or tests positive upon urine drug screen for a substance of abuse.
22. Has a positive pregnancy test at the Screening or Treatment Visit.
23. Has any condition or is taking any medication that would be contraindicated for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in average neuroma foot pain (Diary) with walking using the NPRS | Baseline (mean of Day -7 through Day -1), to week 4 (mean of Day 22 through Day 28)
  Change from Baseline in average neuroma foot pain (Diary) with walking using the NPRS in subjects treated with CNTX-4975 compared with placebo.

SECONDARY OUTCOMES:
Change from Baseline in average neuroma foot pain (Diary) with walking | Baseline (mean of Day -7 through Day -1), Week 1 through Week 12
  Change from Baseline during the Follow-up Period in average neuroma foot pain (Diary) with walking using NPRS (mean of daily pain scores for each week).
Change from Baseline during the Follow-up Period in worst neuroma foot pain (Diary) | Baseline (mean of Day -7 through Day -1),, Week 1 through Week 12
  Change from Baseline during the Follow-up Period in worst neuroma foot pain (Diary) using NPRS (mean of daily pain scores for each week).
Area under the curve (AUC) for average neuroma foot pain (Diary) | Baseline (mean of Day -7 through Day -1), to Week 12
  Area under the curve (AUC) for average neuroma foot pain (Diary) with walking (NPRS).
Foot Function measured by FFI-R-R | Baseline (pre-dose Day 1) to each follow-up visit (Weeks 2, 4, 8, and 12)
  Change from Baseline (pre-dose Day 1) to each follow-up visit (Weeks 2, 4, 8, and 12) in foot function as measured by the FFI-R-R.
QOL as measured by the EQ-5D. | Baseline (pre-dose Day 1) to each follow-up visit (Weeks 2, 4, 8, and 12)
  Change from Baseline (pre-dose Day 1) to each follow-up visit (Weeks 2, 4, 8, and 12) in QOL as measured by the EQ-5D.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Arizona Research Center, Phoenix, Arizona
  - Premier Research, Phoenix, Arizona
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Center for Clinical Research, Inc, Castro Valley, California
  - eStudySite, La Mesa, La Mesa, California
  - TriWest Research Associates, La Mesa, California
  - Chesapeake Research Group, LLC, Pasadena, Maryland
  - Center for Advanced Medicine and Research, City of Saint Peters, Missouri
  - University Orthopedics Center- Altoona, Altoona, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - Allcare Foot and Ankle Center, Arlington, Texas
  - Premier Research, Austin, Texas
  - Endeavor Clinical Trials, PA, San Antonio, Texas
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Jean Brown Research, Salt Lake City, Utah
  - The Education and Research Foundation, Lynchberg, Virginia